CLINICAL TRIAL: NCT05880199
Title: Body Surface Gastric Mapping (BSGM) to Evaluate Patients With Gastrointestinal (GI) Symptoms
Brief Title: BSGM to Evaluate Patients With GI Symptoms
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Auckland, New Zealand (Other)
Responsible Party: Sponsor
Other Study IDs: 21-018520
Record Dates: First submitted 2023-03-24; First posted 2023-05-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Gastrointestinal Motility Disorders in Children; Functional Gastrointestinal Disorders; Gastroparesis; Dyspepsia and Other Specified Disorders of Function of Stomach
Keywords: GI motility; gastroparesis; functional dyspepsia
MeSH Terms: conditions — Gastrointestinal Diseases; Gastroparesis; Dyspepsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Children with functional GI disorders
  Interventions: Device: Body surface gastric mapping device
- Healthy controls
  Interventions: Device: Body surface gastric mapping device

INTERVENTIONS:
Device: Body surface gastric mapping device — A medical device intended to record, store, view and process gastric myoelectrical activity as an aid in the diagnosis of gastrointestinal motility disorders.

SUMMARY:
The goal of this observational study is to learn about gastric myoelectric activity in children with GI symptoms. The main question it aims to answer is which patterns or signals are associated with GI symptoms as measured by a body surface gastric mapping (BSGM) device. Participants will have their stomach activity recorded for up to 4 hours using the BSGM device and log real-time symptoms. Researchers will compare the recordings of healthy children and children with GI symptoms to define abnormal GI patterns.

DETAILED DESCRIPTION:
This is an prospective, multi-cohort study that will focus on adaptation and optimization of a novel non-invasive device called 'Body Surface Gastric Mapping (BSGM)' for use in children including defining and optimizing normal ranges in healthy children, defining abnormal patterns in children with GI symptoms, comparing BSGM patterns with currently used diagnostic tests, and evaluating the mechanisms behind current therapeutic interventions using BSGM patterns as biomarkers.

ELIGIBILITY:
Inclusion Criteria for Cases

1. Males or females age 8 to 25 years.
2. Females ≥11 years of age or who have reached menarche must have a negative urine pregnancy test.
3. Confirmed diagnosis of a Functional Gastrointestinal and/or Motility Disorder OR undergoing one of the following procedures as part of their clinical care at one of the participating centers:

   1. HRVB
   2. PENFS
   3. ADM
   4. Colonic Manometry
   5. Pyloric Botox
   6. Pyloric Dilation
   7. Gastric Scintigraphy
   8. GES
   9. gammaCore
4. Those with a body mass index of < 35.
5. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria for Cases

1. History of skin allergies or a history of extreme sensitivity to cosmetics or lotions. Currently open wounds, abrasions, infected or inflamed abdominal skin. (Please note, majority of feeding tubes can be accommodated by the array placement.)
2. Pregnant women.
3. Those with any condition, where fasting is not recommended by a physician.
4. Any allergies to foods that may be present in the standardized meal that cannot be accommodated with an acceptable substitute meal.
5. Those with physical limitations, who are not able to maintain a relaxed reclined position for the study visit duration.
6. Those with major developmental delay or cognitive impairment, who are not able to report their symptoms/feelings in the questionnaires.
7. Those with GI motility disorders that are limited in the esophagus, and the gastric mapping is restricted to capture relevant data based on the investigator's discretion.
8. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Inclusion Criteria for Controls

1. Males or females age 8 to 25 years.
2. Females ≥11 years of age or who have reached menarche must have a negative urine pregnancy test.
3. Do not have an active Functional Gastrointestinal disorder (FGID) diagnosis and will not be undergoing any procedures outlined in the recruitment plan in the near future.
4. Those with a body mass index of < 35.
5. Individuals may include siblings of those with FGIDs.
6. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria for Controls

1. History of skin allergies or a history of extreme sensitivity to cosmetics or lotions. Currently open wounds, abrasions, infected or inflamed abdominal skin.
2. Pregnant women.
3. Those with any condition, where fasting is not recommended by a physician.
4. Allergies to foods that may be included in the standardized meal that cannot be accommodated with an acceptable substitute meal.
5. Those with physical limitations, who are not able to maintain a relaxed reclined position for the study duration.
6. Those with major developmental delay or cognitive impairment, who are not able to report their symptoms/feelings in the questionnaires.
7. Those with GI motility disorders that are limited in the esophagus, and the gastric mapping is restricted to capture relevant data based on the investigator's discretion.
8. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and adolescents with functional GI and/or motility disorders, and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 685 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
BSGM pediatric reference ranges in healthy controls. | 30 minutes before the meal and 4 hours after having meal.
  Healthy children will be recruited to provide BSGM reference range data. Control data will be used to compute normative data ranges for each key BSGM metric before and after the test meal: slow wave direction, pattern, velocity, frequency, and amplitude.
  For reference ranges:
  * BMI-adjusted amplitude: normal reference range at 5-95% CI
  * Rhythm-Index: normal reference range with cutoff <5% CI
  * Frequency: 5-95% CI
  * Fed: fasted amplitude ratio: <5% CI
  * Slow wave pattern: descriptive
  These outcomes will be measured via the myoelectric activity picked up by the BSGM device.

SECONDARY OUTCOMES:
Abnormal BSGM patterns in participants with functional GI disorders. | 30 minutes before the meal and 4 hours after having meal.
  Abnormal BSGM patterns in participants with GI disorders will be measured by correlating physiological outcomes with symptoms. This will be done by correlating the spectral and spatial data of the stomach collected by the BSGM array with patient symptoms that are entered directly into a symptom-logging app throughout the duration of the BSGM study visit.
Functional disability: Functional disability will be measured by child-reported responses to questions on the Functional Disability Inventory (FDI). | 30 minutes before the meal and 4 hours after having meal.
  The FDI is a validated tool that uses child and parent-reported measure of limitations in children's physical and psychosocial functioning due to their physical health. The instrument consists of 15-items concerning activity limitations during the past two weeks. The four levels of disability are scored as followed: No/Minimal (0-12), Mild (13-20), Moderate (21-29) and Severe (≥30).
Nausea Severity | 30 minutes before the meal and 4 hours after having meal.
  Nausea severity will be assessed by the subject's self-report responses on the Nausea severity scale (NSS) about chronic nausea. The NSS assesses four characteristics of nausea during the past two weeks: number of days with nausea, number of nausea episodes per day, typical nausea duration, and typical intensity of nausea episodes. A total score ranging from 0 - 4 represents the severity of nausea.
Abdominal Pain Severity | 30 minutes before the meal and 4 hours after having meal.
  The correlation of abdominal pain to functional disability will be measured and quantified by the subject's response to the Abdominal Pain Index (API). The API assesses characteristics of abdominal pain during the previous 2 weeks including the number of days with pain, number of pain episodes per day, typical pain episode duration, and typical pain intensity. A total score ranging from 0 (no pain) to - 4 (severe pain) represents the severity of abdominal pain.
Quality of Life - PROMIS-25 Instrument | 30 minutes before the meal and 4 hours after having meal.
  Quality of life will additionally be measured by the participant's completion of the Patient-Reported Outcomes Measurement Information System (PROMIS-25) pediatric profile instrument. The PROMIS-25 is a set of measures from 7 PROMIS domains that evaluate and monitor physical, mental, and social health. This instrument scores questions with a scale from 1 to 5.
Quality of Life - PAGI-QoL | 30 minutes before the meal and 4 hours after having meal.
  Quality of life will additionally be measured by the completion of the Patient Assessment of Upper-GI Disorders Quality of Life (PAGI-QoL) instrument. The PAGI-QoL is a 30-item symptom assessment tool used to assess 6 domains to quantify QoL in adults who have upper GI distress. The PAGI-QoL will be given to subjects aged > 25 years. This instrument scores questions with a scale from 0 to 5.
Quality of life - Pediatric Quality of Life Modules | 30 minutes before the meal and 4 hours after having meal.
  Quality of life and patient reported outcomes will be measured by participants completion of the Pediatric Quality of Life Inventory (PedsQL) and the Pediatric Quality of Life Gastrointestinal Symptom Module Inventory (PedsQL-GI). The PedsQL and PedsQL-GI questionnaires are well-validated measures of child health-related quality of life for children. They are developmentally appropriate, with child self-report and parent-report instruments available for ages 2-25. Scores from each section of these questionnaires are transformed to a 0-100 scale with 0=100 and 4=0. The total score is then calculated by summing all the items over the number of items answered on all the scales.
Compare pediatric BSGM patterns with gastric scintigraphy, a reference diagnostic test. | 30 minutes before the meal and 4 hours after having meal.
  The outcome of the BSGM test, the correlation of the spatial and spectral stomach data with patient symptoms, will be directly compared with the outcomes of each patient that has had a gastric scintigraphy. This will be done by directly comparing the BSGM metrics with the metrics of the gastric scintigraphy (% meal emptied/retained in the stomach, overall clinical assessment of gastric scintigraphy results).
Compare BSGM metrics with the antroduodenal manometry (ADM) metrics. | 30 minutes before the meal and 4 hours after having meal.
  Antoduodenal manometry is a diagnostic test that can be done at the same time as the BSGM study. The data collected by the BSGM study will be directly compared with the sensor data and the ADM for each patient.
Changes in BSGM patterns after heart rate variability biofeedback (HRVB) sessions. | Baseline visit before HRVB and two weeks after HRVB.]
  A BSGM test will be done before and after subjects complete a series of heart rate variability biofeedback (HRVB) sessions. The BSGM patterns will be reviewed for any significant changes that may have been a result of the HRVB sessions.
Changes in BSGM patterns after percutaneous electrical nerve field stimulation (PENFS). | 30 minutes before the meal and 4 hours after having meal.
  A BSGM test will be done before and after subjects have percutaneous electrical nerve field stimulation (PENFS). The BSGM patterns will be reviewed for any significant changes that may have been a result of the PENFS sessions.
Changes in BSGM patterns after pyloric Botulinum toxin (Botox) injection. | 30 minutes before the meal and 4 hours after having meal.
  A BSGM test will be done before and after subjects have pyloric Botulinum toxin (Botox) injections. The BSGM patterns will be reviewed for any significant changes that may have been a result of the pyloric Botox injection.
Changes in BSGM patterns after placement of a gastric electrical stimulator (GES). | 30 minutes before the meal and 4 hours after having meal.
  A BSGM test will be done before GES placement and again while the GES is placed. The BSGM patterns will be reviewed for any significant changes that may be a result of the gastric electrical stimulator.
Compare Colonic Motor Patterns | 1 hour before the meal and 4 hours after having meal.
  The outcome of the colonic BSGM test, the correlation of the spatial and spectral colonic data with patient symptoms, will be directly compared with the outcomes of healthy control subjects through descriptive statistics. An aggregate measure of BSGM will consist of: a stability metric, velocity (mm/s), frequency (cpm), and amplitude (µV).
Correlation Model Parameters | 1 hour before the meal and 4 hours after having meal.
  Colonic BSGM patterns in participants with GI disorders will be correlated with gastrointestinal symptoms that are entered directly into a symptom-logging app throughout the duration of the study visit. Parameters inputted for each patient to this correlation model will include demographics, psychosocial variables (as above), and Colonic BSGM patterns. This model will be reported as an aggregate of demographics, psychosocial variables, and Colonic BSGM patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Hayat Mousa, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (5):
- United States (5):
  - Alliant International University, San Diego, California
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No